CLINICAL TRIAL: NCT05953740
Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of the Long-Acting Injectable of MK-5720 in Participants With Schizophrenia
Brief Title: A Study of MK-5720 in Participants With Schizophrenia (MK-5720-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 5720-001; MK-5720-001 (Other: MSD)
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Saline Solution; Glucose; MK-8189

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Panel A (Experimental): Participants received 7 days of oral MK-8189 4 mg or matched placebo treatment (Period 1), followed by a single intramuscular (IM) injection of MK-5720 35 mg or a dose matched placebo (Period 2).
  Interventions: Drug: MK-5720; Drug: Placebo to MK-5720; Drug: MK-8189; Drug: Placebo to MK-8189
- Panel B (Experimental): Participants received 7 days of oral MK-8189 8 mg or matched placebo treatment (Period 1), followed by a single IM injection of MK-5720 70 mg or a dose matched placebo (Period 2).
  Interventions: Drug: MK-5720; Drug: Placebo to MK-5720; Drug: MK-8189; Drug: Placebo to MK-8189
- Panel C (Experimental): Participants received 7 days of oral MK-8189 up to 16 mg or matched placebo treatment (Period 1), followed by a single IM injection of MK-5720 up to 140 mg or a dose matched placebo (Period 2).
  Interventions: Drug: MK-5720; Drug: Placebo to MK-5720; Drug: MK-8189; Drug: Placebo to MK-8189
- Panel D (Experimental): Participants received 7 days of oral MK-8189 up to 24 mg or matched placebo treatment (Period 1), followed by a single IM injection of MK-5720 up to 280 mg or a dose matched placebo (Period 2).
  Interventions: Drug: MK-5720; Drug: Placebo to MK-5720; Drug: MK-8189; Drug: Placebo to MK-8189
- Panel E (Experimental): Participants received 7 days of oral MK-8189 up to 48 mg or matched placebo treatment (Period 1), followed by a single IM injection of MK-5720 up to 560 mg or a dose matched placebo (Period 2).
  Interventions: Drug: MK-5720; Drug: Placebo to MK-5720; Drug: MK-8189; Drug: Placebo to MK-8189
- Panel F (Experimental): Participants received 7 days of oral MK-8189 up to 48 mg or matched placebo treatment (Period 1), followed by a single IM injection of MK-5720 up to 560 mg or a dose matched placebo (Period 2), after a Pharmacokinetic (PK) break following Panel E.
  Interventions: Drug: MK-5720; Drug: Placebo to MK-5720; Drug: MK-8189; Drug: Placebo to MK-8189

INTERVENTIONS:
Drug: MK-5720 — IM injection
Drug: Placebo to MK-5720 — Placebo IM Injection matched to MK-5720
  Other Names: Normal saline; Dextrose
Drug: MK-8189 — Oral Tablet
Drug: Placebo to MK-8189 — Placebo oral tablet matched to MK-8189

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of single ascending intramuscular doses of MK-5720, and the safety and tolerability of multiple once-daily oral doses of MK-8189, in participants with schizophrenia. The primary study hypothesis is that the administration of MK-5720 is safe and well tolerated.

DETAILED DESCRIPTION:
In Period 1, participants receive once-daily MK-8189 for 7 days, followed by a 72-hour washout. In Period 2, participants receive a single dose of MK-5720.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Meets diagnostic criteria for schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria with the onset of the first episode being no less than 2 years prior to screening and monotherapy with antipsychotics for treatment should be indicated
* Has a history of receiving and tolerating antipsychotics medication within the usual dose range employed for schizophrenia
* Can discontinue the use of all antipsychotic medication at least 5 days or 3 half-lives (which ever in longer) prior to the start of the treatment period and during the study

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Is at imminent risk of self-harm, based on clinical interview and responses on the Columbia-Suicide Severity Rating Scale (C-SSRS), or of harm to others in the opinion of the investigator
* Has history of mental retardation, borderline personality disorder, or organic brain syndrome
* Has a history of neuroleptic malignant syndrome or moderate to severe tardive dyskinesia
* Has a substance-induced psychotic disorder or behavioral disturbance thought to be due to substance abuse
* Has a history of seizure disorder beyond childhood or is receiving treatment with any anticonvulsant to prevent seizures
* Has a family history of sudden death
* Has claustrophobia to a degree that prevents tolerance of magnetic resonance imaging (MRI) scanning procedure
* Has a metallic implant of any sort that prevents MRI examination, or any other contraindication to MRI examination
* Presents any concern by the investigator regarding safe participation in the study or for any other reason the investigator considers the participant inappropriate for participation in the study
* History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food
* Positive test(s) for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV)
* Has received or is currently receiving treatment with clozapine for any length of time
* Has received any live vaccines within 30 days prior to the first dose of study intervention or is scheduled to receive any live vaccine through 60 days following study intervention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - California Clinical Trials Medical Group managed by PAREXEL ( Site 0003), Glendale, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0002), Hallandale, Florida
  - Research Centers of America ( Hollywood ) ( Site 0001), Hollywood, Florida
  - Hassman Research Institute Marlton Site ( Site 0007), Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with schizophrenia were enrolled. Only participants in Panel A, Panel B, and dose-matched placebo were enrolled. Participants were not enrolled in Panels C, D, E, and F and no data was collected.
Groups:
- Panel A: Period 1 MK-8189 4 mg → Period 2 MK-5720 35mg: Participants received 7 days of oral MK-8189 4 mg (Period 1), followed by a single intramuscular (IM) injection of MK-5720 35 mg (Period 2).
- Panel B: Period 1 MK-8189 8 mg → Period 2 MK-5720 70 mg: Participants received 7 days of oral MK-8189 8 mg (Period 1), followed by a single IM injection of MK-5720 70 mg (Period 2).
- Placebo Period 1 → Placebo Period 2: Participants received 7 days of oral MK-8189 dose-matched placebo treatment (Period 1), followed by a single intramuscular (IM) injection of MK-5720 dose-matched placebo treatment (Period 2).
- Panel C: Period 1 MK-8189 16 mg → Period 2 MK-5720 140 mg: Participants received 7 days of oral MK-8189 16 mg (Period 1), followed by a single IM injection of MK-5720 140 mg (Period 2). No participants were enrolled into this arm.
- Panel D: Period 1 MK-8189 24 mg → Period 2 MK-5720 280 mg: Participants received 7 days of oral MK-8189 24 mg (Period 1), followed by a single IM injection of MK-5720 280 mg (Period 2). No participants were enrolled into this arm.
- Panel E: Period 1 MK-8189 48 mg → Period 2 MK-5720 560 mg: Participants received 7 days of oral MK-8189 48 mg (Period 1), followed by a single IM injection of MK-5720 560 mg (Period 2). No participants were enrolled into this arm.
- Panel F: Period 1 MK-8189 48 mg → Period 2 MK-5720 560 mg: Participants received 7 days of oral MK-8189 48 mg (Period 1), followed by a single IM injection of MK-5720 560 mg (Period 2), after a Pharmacokinetic (PK) break following Panel E. No participants were enrolled into this arm.
- Panels C, D, E, and F: Placebo Period 1 → Placebo Period 2: Participants received 7 days of oral MK-8189 dose-matched placebo treatment (Period 1), followed by a single intramuscular (IM) injection of MK-5720 dose-matched placebo (Period 2). No participants were enrolled into this arm.
Period: Period 1
Arm/Group | Panel A: Period 1 MK-8189 4 mg → Period 2 MK-5720 35mg | Panel B: Period 1 MK-8189 8 mg → Period 2 MK-5720 70 mg | Placebo Period 1 → Placebo Period 2 | Panel C: Period 1 MK-8189 16 mg → Period 2 MK-5720 140 mg | Panel D: Period 1 MK-8189 24 mg → Period 2 MK-5720 280 mg | Panel E: Period 1 MK-8189 48 mg → Period 2 MK-5720 560 mg | Panel F: Period 1 MK-8189 48 mg → Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 1 → Placebo Period 2
Started | 6 | 7 | 4 | 0 | 0 | 0 | 0 | 0
Treated | 6 | 7 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 4 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Panel A: Period 1 MK-8189 4 mg → Period 2 MK-5720 35mg | Panel B: Period 1 MK-8189 8 mg → Period 2 MK-5720 70 mg | Placebo Period 1 → Placebo Period 2 | Panel C: Period 1 MK-8189 16 mg → Period 2 MK-5720 140 mg | Panel D: Period 1 MK-8189 24 mg → Period 2 MK-5720 280 mg | Panel E: Period 1 MK-8189 48 mg → Period 2 MK-5720 560 mg | Panel F: Period 1 MK-8189 48 mg → Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 1 → Placebo Period 2
Started | 6 | 6 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 5 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Panels C, D, E, and F were not enrolled, and no data was collected for these panels.
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: Period 1 MK-8189 4 mg → Period 2 MK-5720 35mg | Panel B: Period 1 MK-8189 8 mg → Period 2 MK-5720 70 mg | Placebo Period 1 → Placebo Period 2 | Total
Number analyzed (Participants) | 6 | 7 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (9.4) | 46.3 (11.3) | 51.5 (5.8) | 47.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3
  Male | 6 | 5 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 0 | 4
  Not Hispanic or Latino | 6 | 3 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 3 | 12
  White | 0 | 4 | 1 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience ≥1 Adverse Event (AE) in Period 1
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced one or more AEs is reported here for participants in Period 1. Per protocol, this outcome measure has been reported by panel and dose. As specified by the protocol, Period 2 has been analyzed separately and reported later in the record.
Time Frame: Up to approximately 10 days
Population: All participants in Period 1 who received at least one dose of study treatment and had data available for Period 1. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Panel A: Period 1 MK-8189 4 mg: Participants received 7 days of oral MK-8189 4 mg (Period 1), followed by a single intramuscular (IM) injection of MK-5720 35 mg (Period 2).
- Panel B: Period 1 MK-8189 8 mg: Participants received 7 days of oral MK-8189 8 mg (Period 1), followed by a single IM injection of MK-5720 70 mg (Period 2).
- Placebo Period 1: Participants received 7 days of oral MK-8189 dose-matched placebo treatment (Period 1), followed by a single intramuscular (IM) injection of MK-5720 dose-matched placebo treatment (Period 2).
- Panel C: Period 1 MK-8189 16 mg: Participants received 7 days of oral MK-8189 16 mg (Period 1), followed by a single IM injection of MK-5720 140 mg (Period 2). No participants were enrolled into this arm.
- Panel D: Period 1 MK-8189 24 mg: Participants received 7 days of oral MK-8189 24 mg (Period 1), followed by a single IM injection of MK-5720 280 mg (Period 2). No participants were enrolled into this arm.
- Panel E: Period 1 MK-8189 48 mg: Participants received 7 days of oral MK-8189 48 mg (Period 1), followed by a single IM injection of MK-5720 560 mg (Period 2). No participants were enrolled into this arm.
- Panel F: Period 1 MK-8189 48 mg: Participants received 7 days of oral MK-8189 48 mg (Period 1), followed by a single IM injection of MK-5720 560 mg (Period 2), after a Pharmacokinetic (PK) break following Panel E. No participants were enrolled into this arm.
- Panels C, D, E, and F: Placebo Period 1: Participants received 7 days of oral MK-8189 dose-matched placebo treatment (Period 1), followed by a single intramuscular (IM) injection of MK-5720 dose-matched placebo (Period 2). No participants were enrolled into this arm.
Arm/Group | Panel A: Period 1 MK-8189 4 mg | Panel B: Period 1 MK-8189 8 mg | Placebo Period 1 | Panel C: Period 1 MK-8189 16 mg | Panel D: Period 1 MK-8189 24 mg | Panel E: Period 1 MK-8189 48 mg | Panel F: Period 1 MK-8189 48 mg | Panels C, D, E, and F: Placebo Period 1
Number analyzed (Participants) | 6 | 7 | 4 | 0 | 0 | 0 | 0 | 0
Participants | 1 | 4 | 2 |  |  |  |  |

2. Primary Outcome: Number of Participants Who Experience ≥1 AE(s) in Period 2
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced one or more AEs is reported here for participants in Period 2. Per protocol, this outcome measure has been reported by panel and dose. As specified by the protocol, Period 1 has been analyzed separately and reported earlier in the record.
Time Frame: Up to approximately 72 days
Population: All participants in Period 2 who received at least one dose of study treatment and had data available for Period 2. In Panel B 1 participant discontinued treatment between Period 1 and Period 2. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Panel A: Period 2 MK-5720 35mg: Participants received 7 days of oral MK-8189 4 mg (Period 1), followed by a single intramuscular (IM) injection of MK-5720 35 mg (Period 2).
- Panel B: Period 2 MK-5720 70 mg: Participants received 7 days of oral MK-8189 8 mg (Period 1), followed by a single IM injection of MK-5720 70 mg (Period 2).
- Placebo Period 2: Participants received 7 days of oral MK-8189 dose-matched placebo treatment (Period 1), followed by a single intramuscular (IM) injection of MK-5720 dose-matched placebo treatment (Period 2).
- Panel C: Period 2 MK-5720 140 mg: Participants received 7 days of oral MK-8189 16 mg (Period 1), followed by a single IM injection of MK-5720 140 mg (Period 2). No participants were enrolled into this arm.
- Panel D: Period 2 MK-5720 280 mg: Participants received 7 days of oral MK-8189 24 mg (Period 1), followed by a single IM injection of MK-5720 280 mg (Period 2). No participants were enrolled into this arm.
- Panel E: Period 2 MK-5720 560 mg: Participants received 7 days of oral MK-8189 48 mg (Period 1), followed by a single IM injection of MK-5720 560 mg (Period 2). No participants were enrolled into this arm.
- Panel F: Period 2 MK-5720 560 mg: Participants received 7 days of oral MK-8189 48 mg (Period 1), followed by a single IM injection of MK-5720 560 mg (Period 2), after a Pharmacokinetic (PK) break following Panel E. No participants were enrolled into this arm.
- Panels C, D, E, and F: Placebo Period 2: Participants received 7 days of oral MK-8189 dose-matched placebo treatment (Period 1), followed by a single intramuscular (IM) injection of MK-5720 dose-matched placebo (Period 2). No participants were enrolled into this arm.
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 6 | 6 | 4 | 0 | 0 | 0 | 0 | 0
Participants | 1 | 2 | 1 |  |  |  |  |

3. Primary Outcome: Number of Participants Who Discontinue Study Due to an AE in Period 1
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment due to an AE is reported here for participants in Period 1. Per protocol, this outcome measure has been reported by panel and dose. As specified by the protocol, Period 2 has been analyzed separately and reported later in the record.
Time Frame: Up to approximately 10 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Period 1 MK-8189 4 mg | Panel B: Period 1 MK-8189 8 mg | Placebo Period 1 | Panel C: Period 1 MK-8189 16 mg | Panel D: Period 1 MK-8189 24 mg | Panel E: Period 1 MK-8189 48 mg | Panel F: Period 1 MK-8189 48 mg | Panels C, D, E, and F: Placebo Period 1
Number analyzed (Participants) | 6 | 7 | 4 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 1 | 0 |  |  |  |  |

4. Primary Outcome: Number of Participants Who Discontinue Study Due to an AE in Period 2
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment due to an AE is reported here for participants in Period 2. Per protocol, this outcome measure has been reported by panel and dose. As specified by the protocol, Period 1 has been analyzed separately and reported earlier in the record.
Time Frame: Up to approximately 72 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 6 | 6 | 4 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 0 |  |  |  |  |

5. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Last Quantifiable Concentration (AUC0-last) of MK-5720
Description: AUC0-last was defined as the area under the concentration-time curve from time zero to time of last measurable concentration of MK-5720. Blood samples were collected at specified intervals were used to estimate AUC0-last following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 24, 48, 96, 120, 144, 168, 192, 216, 264, 288, 312, 336, 360, 384, 432, 456, 504, 672, 840, 1008, 1176, and 1320 hours postdose
Population: Per protocol population includes all participants who complied with the protocol, had received MK-8189 treatment in Period 1 and MK-5720 treatment in Period 2, and had data available. Per protocol, placebo arms were not included in any PK outcome analyses. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr*nM | 34.3 (128.3) | 73.3 (96.2) |  |  |  |  |  |

6. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC-inf) of MK-5720
Description: AUC0-inf is defined as the area under concentration-time curve of MK-5720 from time zero to infinity. Blood samples were collected at specified intervals for the determination of AUC-inf following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr*nM | 70.0 (61.6) | 134 (61.6) |  |  |  |  |  |

7. Primary Outcome: Maximum Serum Concentration (Cmax) of MK-5720
Description: Cmax is defined as the maximum concentration of MK-5720 reached. Blood samples were collected at specified intervals for the determination of Cmax following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
nM | 0.165 (156.2) | 0.473 (105.1) |  |  |  |  |  |

8. Primary Outcome: Time to Maximum Concentration (Tmax) of MK-5720
Description: Tmax is defined as the time to maximum concentration of MK-5720 reached. Blood samples were collected at specified intervals for the determination of Tmax following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr | 48.00 [0.50 to 96.00] | 108.00 [4.00 to 192.12] |  |  |  |  |  |

9. Primary Outcome: Apparent Clearance (CL/F) of MK-5720
Description: CL/F is the rate at which the MK-5720 is completely removed from plasma. Blood samples were collected at specified intervals for the determination of CL/F following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hr
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Liters/hr | 892 (61.6) | 933 (61.6) |  |  |  |  |  |

10. Primary Outcome: Apparent Volume of Distribution (Vz/F) of MK-5720
Description: Vz/F is the apparent volume of distribution of MK-5720. Blood samples were collected at specified intervals for the determination of Vz/F following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Liters | 55400 (83.2) | 218000 (243.8) |  |  |  |  |  |

11. Primary Outcome: Apparent Terminal Half-life (t1/2) of MK-5720
Description: t1/2 is defined as the time required to divide plasma concentration of MK-5720 by half after reaching pseudo-equilibrium. Blood samples were collected at specified intervals for the determination t1/2 following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr | 43.0 (15.9) | 162 (271.2) |  |  |  |  |  |

12. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to 28 Days (AUC0-28d) of MK-8189
Description: AUC0-28d is defined as the area under the concentration-time curve from time zero to 28 days of MK-8189 (a metabolite of MK-5720). Blood samples were collected at specified intervals for the determination of AUC0-28d for MK-8189 following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 24, 48, 96, 120, 144, 168, 192, 216, 264, 288, 312, 336, 360, 384, 432, 456, 504, and 672 hours postdose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr*nM | 2850 (4121.1) | 29800 (89.3) |  |  |  |  |  |

13. Primary Outcome: AUC0-inf of MK-8189
Description: AUC0-inf is defined as the area under concentration-time curve from time zero to infinity of MK-8189 (a metabolite of MK-5720). Blood samples were collected at specified intervals for the determination of AUC0-inf for MK-8198 following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr*nM | 8400 (75.3) | 31900 (93.9) |  |  |  |  |  |

14. Primary Outcome: Cmax of MK-8189
Description: Cmax is defined as the maximum concentration of MK-8189 (a metabolite of MK-5720) reached. Blood samples were collected at specified intervals for the determination of Cmax for MK-8198 following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
nM | 18.8 (569.7) | 104 (90.1) |  |  |  |  |  |

15. Primary Outcome: Tmax of MK-8189
Description: Tmax is defined as the time to maximum concentration of MK-8189 (a metabolite of MK-5720). Blood samples were collected at specified intervals for the determination of Tmax for MK-8198 following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr | 96.00 [24.00 to 504.00] | 120.00 [96.00 to 288.00] |  |  |  |  |  |

16. Primary Outcome: Concentration at Day 28 (C28d) of MK-8189
Description: C28d is defined as the maximum concentration from time zero to 28 days of MK-8189 (a metabolite of MK-5720). Blood samples were collected at specified intervals for the determination of C28d for MK-8198 following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose. In cases where C28d values were below the limit of quantitation, geometric mean was not calculable and indicated as "NA."
Time Frame: as for outcome 12
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
nM | NA (NA) — NA = Geometric mean (% GCV) were not calculable as plasma concentrations were the below the limit of quantitation. | 2.96 (693.7) |  |  |  |  |  |

17. Primary Outcome: CL/F of MK-8189
Description: CL/F is the rate at which the MK-8189 (a metabolite of MK-5720) is completely removed from plasma. Blood samples were collected at specified intervals for the determination of CL/F for MK-8198 following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hr
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Liters/hr | 7.43 (75.3) | 3.92 (93.9) |  |  |  |  |  |

18. Primary Outcome: Vz/F of MK-8189
Description: Vz/F is the apparent volume of distribution of MK-8189 (a metabolite of MK-5720). Blood samples were collected at specified intervals for the determination of Vz/F for MK-8198 following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Liters | 697 (97.0) | 593 (126.7) |  |  |  |  |  |

19. Primary Outcome: t1/2 of MK-8189
Description: t1/2 is defined as the time required to divide plasma concentration of MK-8189 (a metabolite of MK-5720) by half after reaching pseudo-equilibrium. Blood samples were collected at specified intervals for the determination of Half-life (t1/2) for MK-8198 following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure has been reported by panel and dose.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr | 65.0 (62.5) | 105 (71.3) |  |  |  |  |  |

20. Secondary Outcome: Panels D, E, and F: C28d Tied to Specific Exposures of MK-8189
Description: C28d tied to specific exposures of MK-8189 is defined as the maximum concentration from time zero to 28 days of MK-8189 tied to specific exposures. Blood samples were collected at specified intervals for the determination of C28d tied to specific exposures of MK-8189 (metabolite of MK-5720) following a single dose administration of MK-5720 in Period 2. Per protocol, this outcome measure is specific for Panels D, E, and F only. Panels C, D, E and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 24, 48, 96, 120, 144, 168, 192, 216, 264, 288, 312, 336, 360, 384, 432, 456, 504, and 672 postdose
Population: Per protocol, this outcome measure is specific for Panels D, E, and F only. Panels C, D, E and F were not enrolled, and no data was collected for this outcome measure. Per protocol, placebo arms were not included in any PK outcome analyses.
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Panels C, D, E, and F: AUC0-28d of MK-8189 in Gluteal Muscle Versus AUC0-28 of MK-8189 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of AUC0-28 of MK-8189 (a metabolite of MK-5720) after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. AUC0-28 is defined as the area under the plasma concentration-time curve from time zero to 28 days of MK-8189. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 12
Population: Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A and B. Per protocol, placebo arms were not included in any PK outcome analyses. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Panels C, D, E, and F: AUC0-inf of MK-8189 in Gluteal Muscle Versus AUC0-inf of MK-8189 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of AUC-inf of MK-8189 (a metabolite of MK-5720) after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. AUC0-inf is defined as the area under concentration-time curve from time zero to infinity of MK-8189. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Panels C, D, E, and F: Cmax of MK-8189 in Gluteal Muscle Versus Cmax of MK-8189 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of Cmax of MK-8189 (a metabolite of MK-5720) after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. Cmax is defined as the maximum concentration of MK-8189. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Panels C, D, E, and F: Tmax of MK-8189 in Gluteal Muscle Versus Tmax of MK-8189 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for determination of Tmax of MK-8189 (a metabolite of MK-5720) after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. Tmax is defined as the time to maximum concentration of MK-8189. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 24, 48, 96, 120, 144, 168, 192, 216, 264, 288, 312, 336, 360, 384, 432, 456, 504, 672, 840, 1008, 1176, 1320 hours postdose
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Panels C, D, E, and F: C28d of MK-8189 in Gluteal Muscle Versus C28d in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of C28d of MK-8189 (a metabolite of MK-5720) after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. C28d is defined as the maximum concentration from time zero to 28 days of MK-8189. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 12
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Panels C, D, E, and F: CL/F of MK-8189 in Gluteal Muscle Versus CL/F in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of CL/F of MK-8189 (a metabolite of MK-5720) after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. CL/F is the rate at which the MK-8189 is completely removed from plasma. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Panels C, D, E, and F: Vz/F of MK-8189 in Gluteal Muscle Versus Vz/F of MK-8189 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of distribution of MK-8189 (metabolite of MK-5720) after administration of MK-5720 (Period 2) in the gluteal muscle versus deltoid muscle. Vz/F is the apparent volume of distribution of MK-8189. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Panels C, D, E, and F: t1/2 of MK-8189 in Gluteal Muscle Versus t1/2 of MK-8189 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of t1/2 of MK-8189 (metabolite of MK-5720) after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. t1/2 is defined as the time required divide plasma concentration of MK-8189 (metabolite of MK-5720) by half after reaching pseudo-equilibrium. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Panels C, D, E, and F: AUC0-last of MK 5720 in Gluteal Muscle Versus AUC0-last of MK-5720 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of AUC0-last after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. AUC0-last is defined as the area under the concentration-time curve from time zero to time of last measurable concentration of MK-5720. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Panels C, D, E, and F: AUC0-inf of MK-5720 in Gluteal Muscle Versus AUC0-inf of MK-5720 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of AUC-inf after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. AUC0-inf is defined as the area under concentration-time curve from time zero to infinity. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Panels C, D, E, and F: Cmax of MK-5720 in Gluteal Muscle Versus Cmax of MK-5720 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of Cmax after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. Cmax is defined as the maximum concentration of MK-5720 reached. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Panels C, D, E, and F: Tmax of MK-5720 in Gluteal Muscle Versus Tmax of MK-5720 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of Tmax after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. Tmax is defined as the time to maximum concentration of MK-5720 reached. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Panels C, D, E, and F: CL/F of MK-5720 in Gluteal Muscle Versus CL/F of MK-5720 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination of CL/F after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. CL/F is the rate at which the MK-5720 is completely removed from plasma. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

34. Secondary Outcome: Panels C, D, E, and F: Vz/F of MK-5720 in Gluteal Muscle Versus Vz/F of MK-5720 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination Vz/F after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. Vz/F is the apparent volume of distribution of MK-5720. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Panels C, D, E, and F: t1/2 of MK-5720 in Gluteal Muscle Versus t1/2 of MK-5720 in Deltoid Muscle
Description: Blood samples were to be collected at specified intervals for the determination t1/2 after administration of MK-5720 (Period 2) in the gluteal muscle and deltoid muscle. t1/2 is defined as the time required to divide plasma concentration of MK-5720 by half after reaching pseudo-equilibrium. Per protocol, this outcome measure is specific for Panels C, D, E, and F, and data was not planned or collected for Panels A or B. Panels C, D, E, and F were not enrolled, and no data was collected for this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 21
Arm/Group | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2 | Panel C: Period 2 MK-5720 140 mg | Panel D: Period 2 MK-5720 280 mg | Panel E: Period 2 MK-5720 560 mg | Panel F: Period 2 MK-5720 560 mg | Panels C, D, E, and F: Placebo Period 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 82 days
Description: Population for All-cause mortality was All Randomized Participants. Population for non-serious adverse events and serious adverse events consists of all randomized participants who received at least 1 dose of the study intervention and have provided safety data at any time during the study. Panels C, D, E, and F were not enrolled, and no data was collected for these panels.
Arm/Group | Panel A: Period 1 MK-8189 4 mg | Panel B: Period 1 MK-8189 8 mg | Placebo Period 1 | Panel A: Period 2 MK-5720 35mg | Panel B: Period 2 MK-5720 70 mg | Placebo Period 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/4 | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/4 | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 4/7 | 2/4 | 1/6 | 2/6 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: Period 1 MK-8189 4 mg (N=6) | Panel B: Period 1 MK-8189 8 mg (N=7) | Placebo Period 1 (N=4) | Panel A: Period 2 MK-5720 35mg (N=6) | Panel B: Period 2 MK-5720 70 mg (N=6) | Placebo Period 2 (N=4)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT05953740/Prot_SAP_000.pdf